CLINICAL TRIAL: NCT01347554
Title: Comparison of the Efficacy of Everolimus-Eluting Versus Zotarolimus-Eluting Stent for Coronary Lesions in Acute Myocardial Infarction
Brief Title: Efficacy of Everolimus-Eluting Versus Zotarolimus-Eluting Sten for Coronary Lesions in Acute Myocardial Infarction
Acronym: EVERZOTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVZT_2.0
Record Dates: First submitted 2011-04-27; First posted 2011-05-04 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction
Keywords: drug-eluting stent; everolimus; zotarolimus; myocardial ischemia; cardiovascular diseases; MACE; safety
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xience V stent group (Active Comparator): Xience V (Everolimus eluting stent) insertion in patients with acute myocardial infarction
  Interventions: Device: Everolimus eluting stent
- Endeavor resolute group (Active Comparator): Endeavor resolute (Zotarolimus eluting stent) insertion in patients with acute myocardial infarction
  Interventions: Device: Zotarolimus eluting stent

INTERVENTIONS:
Device: Everolimus eluting stent — Comparison of the safety and efficacy between everolimus-eluting stent and zotarolimus-eluting stent resolute
  Other Names: Xience V; Promus or Promus element
  Arms: Xience V stent group
Device: Zotarolimus eluting stent — Comparison of the safety and efficacy between everolimus-eluting stent and zotarolimus-eluting stent resolute
  Other Names: Endeavor resolute
  Arms: Endeavor resolute group

SUMMARY:
Most of the previous data regarding the efficacy of the everolimus-eluting stent (EES) was derived from studies comparing EES with bare metal stent (BMS) or EES with paclitaxel-eluting (PES). Although sirolimus-eluting stents (SES) have been shown to be the most efficacious drug regarding inhibition of neointima and late loss, there have been no previous head to head comparisons between EES and zotarolimus-eluting stent (ZES). Both everolimus and sirolimus are macrocyclic lactones that target the mTOR (mammalian target of rapamycin) to reduce vascular smooth muscle proliferation after vessel injury and therefore in principle may show similar results after stenting in humans. Data pooled from the EES arm that received follow up angiography in the SPIRIT III trial and the SES arm in the SIRIUS trial show similar rates of binary restenosis and late loss. However, the stent and polymer platform is not the same between the EES and ZES and it is reported that the EES system has the thinnest stent + polymer thickness (88.6um) of all of the previously KFDA-approved drug-eluting stent (DES). In addition, there are no data available on the efficacy of the EES and ZES in "real world" lesions other than the selected lesions studied in the previous trials, such as acute myocardial infarction.

DETAILED DESCRIPTION:
Previous randomized trials have shown the efficacy of a slow-release polymeric sirolimus-eluting stent (CYPHER, Cordis, Warren, NJ, USA), paclitaxel-eluting stent (TAXUS, Boston Scientific, Natick, MA, USA), and zotarolimus-eluting stent (Endeavor, Medtronic, Minneapolis, MN, USA) over bare metal stents in reducing neointimal hyperplasia, late luminal loss, and angiographic restenosis leading to decreased target lesion revascularization. The everolimus-eluting stent (XIENCE V, Abott Vascular, Santa Clara, CA, USA, PROMUS, Boston Scientific, Natick, MA, USA) is a newly developed drug eluting stent using the MULTILINK VISION® stent platform combined with the drug everolimus contained in a polymer coating.

In the first-in-man SPIRIT First clinical trial, XIENCE V showed a significant benefit over the bare metal VISION stent. Compared with late loss of 0.85 ± 0.36mm in the VISION arm, XIENCE V reduced late loss by 88% (0.10 ± 0.23mm). Also the clinical safety of XIENCE V was confirmed with a 6-month MACE rate of 7.7%. In the SPIRIT II clinical trial, which compared the efficacy and safety of the XIENCE V stent versus the TAXUS PECSS stent, the primary endpoint was met showing a non-inferiority of the XIENCE V compared with the TAXUS regarding in-stent late loss at 180 days. Actually, XIENCE V was superior to TAXUS and reduced in-stent late loss by 72% from a mean of 0.36 mm to 0.11 mm. In addition, analysis of other key clinical endpoints showed a lower rate of ischemia driven MACE (2.7% vs. 6.5% for XIENCE V vs. TAXUS) and protocol-defined stent thrombosis (0.5% vs. 1.3% for XIENCE V vs. TAXUS). The lower rate of ischemia driven MACE at 180 days was sustained through 1 year and there were no new instances of late stent thrombosis in either group up to 1 year.

The SPIRIT III RCT was a prospective, 2:1 randomized, active-controlled, single blinded, parallel, multi-center clinical evaluation of the XIENCE V Everolimus Eluting Coronary Stent System (XIENCE V EECSS) compared to TAXUS Paclitaxel Eluting Coronary Stent System (TAXUS PECSS) in the treatment of up to two de novo lesions. This pivotal clinical trial was designed to demonstrate the non-inferiority of the XIENCE V EECSS to the TAXUS PECSS. Patients were randomized 2:1 to XIENCE V or TAXUS and the primary endpoint was in-segment late loss at 240 days. The results showed a mean in-segment late loss of 0.14mm for XIENCE V and 0.28 mm for TAXUS (p<0.001 for non-inferiority, p=0.0037 for superiority). The secondary endpoint, which was ischemia-driven target vessel failure (TVF), was 7.6% for XIENCE V and 9.7% for TAXUS, confirming the non-inferiority of XIENCE V. Furthermore, the rate of definite and probable stent thrombosis was 1.1% and 0.6% for XIENCE V and TAXUS, respectively.

With a recent approval of new DES, zotarolimus-eluting stent (Endeavor, Medtronic, Minneapolis, MN), other comparison studies have been conducted to compare Endeavor zotarolimus-eluting stent with the sirolimus-eluting stent and paclitaxel-eluting stent. zotarolimus and sirolimus share some common structural and biological properties. In vitro data suggest that sirolimus and tetrazole containing rapamycin analogs have similar inhibitory effects in a mixed lymphocyte reaction assay. The ENDEAVOR clinical trials are currently in progress to evaluate a phosphoryl choline (PC)-coated zotarolimus-eluting stent(ZES) for the prevention of restenosis. The Endeavor zotarolimus-eluting stent utilizes a cobalt alloy balloon-expandable stent (Driver; Medtronic) with a geometry similar to the stainless steel stent used in this preliminary study (S7; Medtronic). The Endeavor ZES also employees a PC strut surface coating as the drug delivery reservoir with a dose of 10 g/mm of ABT-578. The Endeavor (ZES), however, differs from the stent used in this experimental study by the addition of a drug-free PC topcoat to serve as a diffusion barrier to retard drug release from the polymer reservoir. Angiographic analysis at 4 months in the 100-patient focal de novo lesion ENDEAVOR I feasibility study demonstrated a mean in-stent percent diameter stenosis of approximately 14% and a late lumen loss of 0.3 mm with a low frequency of target lesion revascularization (1%). The clinical outcomes from the ENDEAVOR II (1,500 patients randomized to ABT-578 or bare metal stent) and the ENDEAVOR III (436 patients randomized 3:1 to ABT-578 or Cypher) trials as well as other ongoing studies showed efficacy of the PC-coated ABT-578-eluting stent. In ENDEAVOR III study, the Endeavor stent had larger late loss and higher binary restenosis in both the analysis segment and stented segment.

Most of the previous data regarding the efficacy of the EES was derived from studies comparing EES with BMS or EES with PES. Although sirolimus eluting stents (SES) have been shown to be the most efficacious drug eluting stent regarding inhibition of neointima and late loss, there have been no previous head to head comparisons between EES and ZES. Both everolimus and sirolimus are macrocyclic lactones that target the mTOR (mammalian target of rapamycin) to reduce vascular smooth muscle proliferation after vessel injury and therefore in principle may show similar results after stenting in humans. Data pooled from the EES arm that received follow up angiography in the SPIRIT III trial and the SES arm in the SIRIUS trial show similar rates of binary restenosis and late loss. However, the stent and polymer platform is not the same between the EES and ZES and it is reported that the EES system has the thinnest stent + polymer thickness (88.6um) of all of the previously KFDA-approved DES. In addition, there are no data available on the efficacy of the EES and ZES in "real world" lesions other than the selected lesions studied in the previous trials, such as acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Chest pain duration more than 10 minutes
* At least on of the following criteria
* A. ECG change (T inversion, ST depression or ST elevation)
* B. Cardiac enzyme elevation more than upper normal limit
* Significant coronary artery stenosis (>50% by visual estimate)
* The patient or guardian agrees to the study

Exclusion Criteria:

* Stent thrombosis
* Left main disease
* Cardiogenic shock
* Cronic kidney disease or renal failure requiring hemodialysis
* History of bleeding diathesis or known coagulopathy
* Gastrointestinal or genitourinary bleeding within the prior 3 months
* History of major surgery within 2 months
* Planned surgery requiring cessation of clopidogrel within 12 months of percutaneous coronary intervention (PCI)
* Serious patients whose life expectancy <1 year or severe infectious status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hwan Lee, MD, PhD, Principal Investigator — Division of Cardiology, Department of Internal Medicine, Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital
Locations (1):
- Yonsei University Wonju College of Medicine; Wonju Severance Christian Hospital, Wŏnju, South Korea

REFERENCES:
- [Derived] Ahn SG, Choi HH, Lee JH, Lee JW, Youn YJ, Yoo SY, Cho BR, Lee SH, Yoon J. The impact of initial and residual thrombus burden on the no-reflow phenomenon in patients with ST-segment elevation myocardial infarction. Coron Artery Dis. 2015 May;26(3):245-53. doi: 10.1097/MCA.0000000000000197. PMID 25503419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2009 and December 2010, we undertook a multicenter, prospective, randomized trial in 4 tertiary university hospitals.
Pre-assignment Details: Patients with acute myocardial infarction were eligible if they had at least one lesion with a diameter stenosis of 50%or more. Before randomization, 3 patients withdrew consent and 18 patients did not meet inclusion criteria among 500 patients.
Period: Overall Study
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Started | 237 | 242
Completed | 230 (Final TIMI flow grade 0 or 1 patients or failed PCI cases (N=7) were excluded.) | 231 (Final TIMI flow grade 0 or 1 patients or failed PCI cases (N=11) were excluded.)
Not Completed | 7 | 11
Not completed — Lack of Efficacy | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xience V Stent Group | Endeavor Resolute Group | Total
Number analyzed (Participants) | 230 | 231 | 461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 106 | 212
  >=65 years | 124 | 125 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (12.8) | 64.5 (11.8) | 64.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 62 | 125
  Male | 167 | 169 | 336
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 230 | 231 | 461

OUTCOME MEASURES:

1. Primary Outcome: Device-oriented Composite Outcome
Description: defined as a composite of cardiac death, Myocardial infarction not clearly attributable to a nontarget vessel and target lesion revascularization
Time Frame: Two year
Measure: Number; unit: participants
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Number analyzed (Participants) | 230 | 231
participants | 12 | 13

2. Secondary Outcome: Device-oriented Composite Outcome
Description: defined as a composite of all-cause mortality, any MI (includes non-target vessel territory) and repeat revascularization (includes all target and non-target vessel)
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Number analyzed (Participants) | 230 | 231
participants | 20 | 24

3. Secondary Outcome: Stent Thrombosis
Description: Definite and probable stent thrombosis
Time Frame: Two years
Measure: Number; unit: participants
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Number analyzed (Participants) | 230 | 231
participants | 0 | 7

4. Secondary Outcome: Any Bleeding
Time Frame: Two year
Measure: Number; unit: participants
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Number analyzed (Participants) | 230 | 231
participants | 7 | 11

ADVERSE EVENTS:
Time Frame: Two year
Arm/Group | Xience V Stent Group | Endeavor Resolute Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Relatively small number of sample size. Therefore, our result may be underpowerd. The incidence of clinical events were low. And we did not record the compliance of dual antiplatelet therapy for at least 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No